CLINICAL TRIAL: NCT06307496
Title: Video Interventions for Dependence On Smoking (VIDeOS) for Cancer Patients: A Randomized Controlled Pilot Study
Brief Title: VIDeOS for Smoking Cessation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Kinsey Pebley, Post Doctoral-Fellow, Medical University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: Pro00133913
Record Dates: First submitted 2024-03-05; First posted 2024-03-12 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Cancer; Smoking Cessation
Keywords: Videos
MeSH Terms: conditions — Neoplasms; Smoking Cessation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Videos (Experimental): Participants will be sent links to smoking cessation videos to watch.
  Interventions: Other: Smoking cessation intervention
- NCI Pamphlet (Active Comparator): Participants will be sent links to NCI's "Clearing the Air" to read.
  Interventions: Other: Informational intervention

INTERVENTIONS:
Other: Smoking cessation intervention — Receive links to smoking cessation videos
  Arms: Videos
Other: Informational intervention — Receive NCI's "Clearing the Air" booklet
  Arms: NCI Pamphlet

SUMMARY:
The purpose of the current study is to pilot the efficacy, feasibility, and acceptability of an evidence-based smoking cessation intervention adapted for cancer patients and delivered via video. Investigators aim to assess if this intervention is considered acceptable by participants, feasible to implement, and effective at increasing knowledge about smoking cessation before conducting a fully powered clinical trial.

DETAILED DESCRIPTION:
A randomized controlled pilot study is being conducted to test the acceptability and feasibility of a smoking cessation intervention tailored for cancer patients that is delivered via video. Participants will be in a video intervention or control group that receives information about quitting smoking. Participants will complete surveys prior to randomization, and will complete additional surveys one week, one month, and three months post-randomization to provide their thoughts about the videos, information about changes to smoking behaviors, and knowledge about quitting smoking.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* Diagnosed with cancer (any type)
* Receiving care at Medical University of South Carolina
* Reads and understands English language
* Currently smoking cigarettes (any amount)

Exclusion Criteria:

- Unstable or poorly managed medical or psychiatric conditions that impair cognition and ability to provide informed consent (e.g., dementia, active psychosis).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2024-09-24 (Actual); Primary Completion 2025-09-10 (Actual); Study Completion 2025-09-10 (Actual)

PRIMARY OUTCOMES:
Acceptability | 1 week post-randomization
  Acceptability will be measured using the Acceptability of Intervention measure, which contains four items with answer options on a scale from 1-5, with higher scores indicating higher acceptability. We will consider the intervention "acceptable" if an average score of 4 or higher is obtained.
Feasibility | 1 week post-randomization
  Feasibility will be measured using the Feasibility of Intervention measure, which contains four items with answer options on a scale from 1-5, with higher scores indicating higher feasibility. We will consider the intervention "feasible" if an average score of 4 or higher is obtained.
Retention Rates | 1 week, 1 month, and 3 months post-randomization
  We will determine if there are differences in retention rates between intervention groups.

SECONDARY OUTCOMES:
Changes in knowledge about quitting smoking | Baseline, 1 week, 1 month, and 3 months post-randomization
  We will assess changes in knowledge about tools to quit smoking and the role of nicotine, etc. from prior to randomization (before the intervention is delivered) to post-randomization follow-ups. These questions will be generated by the study investigators based on video content.
Changes in smoking behaviors | 1 week, 1 month, and 3 months post-randomization
  We will assess the number of 24-hour quit attempts and 7-day point prevalence at 1 week, 1 month, and 3 month follow-ups.

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

DOCUMENTS (1):
  • Informed Consent Form (2024-07-11): https://cdn.clinicaltrials.gov/large-docs/96/NCT06307496/ICF_000.pdf